CLINICAL TRIAL: NCT02785536
Title: RITCH: Reducing Disparities in Tobacco Cessation Outcomes
Acronym: RITCh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The City College of New York (Other)
Collaborators: Virginia Tech Carilion School of Medicine and Research Institute (Other)
Responsible Party: Principal Investigator, Christine Sheffer, Associate Professor, The City College of New York
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #361627
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Smoking Cessation
Keywords: minority health; social class; healthcare disparities; tobacco use disorder
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Treatment (Active Comparator): The standard treatment was a well-established, manual-driven, multicomponent CBT for tobacco dependence that has been delivered in multiple modalities (i.e., group, individual, and telephone), used in numerous studies, and considered intensive, comprehensive, and consistent with the Public Health Service Clinical Practice Guideline.
  Interventions: Behavioral: Standard Treatment
- RITCh Treatment (Experimental): The RITCh treatment is an adaptation of the standard treatment which proactively addresses the needs and experiences of a diverse group of lower SES smokers as well as ensures that the treatment is culturally congruent and experientially resonant for African Americans while maintaining the same amount of treatment contact (i.e., six one-hour sessions).
  Interventions: Behavioral: RITCh Treatment

INTERVENTIONS:
Behavioral: RITCh Treatment — The RITCh treatment increased the emphasis on stress management, negative affect management and utilized language and activities to foster an internal locus of control. Activities were added to address impulsive decision-making, develop home smoking policies, increase the positive valance of treatment, and address barriers to use of the nicotine patches. The treatment materials were also tailored with numerous examples relevant to lower SES groups and African Americans. For example: stress management components specifically address financial stress, discrimination, and micro-aggressions; treatment utilization components include reinforcing the value of individual contributions to the group, structured positive feedback among group members at every session, sending "missed you" post cards signed by all group members to participants who miss a treatment session, specifically addressing myths about nicotine patch use, and practicing the application of nicotine patches together.
  Arms: RITCh Treatment
Behavioral: Standard Treatment — The components of the standard treatment include education and activities in which participants gain an understanding of the biopsychosocial underpinnings of tobacco dependence and the cue-urge-response cycle of smoking. Interventions include self-monitoring, guided scheduled rate reduction, treatment goal setting, medication education, stress management, cognitive and behavioral strategies for managing cravings and cues, problem-solving, conflict management, enhancing social support, relapse prevention, and cigarette refusal training. A participant workbook was provided that corresponded to the activities in the treatment sessions.
  Arms: Standard Treatment

SUMMARY:
Tobacco use is a leading contributor to racial and socioeconomic health disparities in the US primarily due to an unequal burden of tobacco-related disease from a disproportionate share of smokers in African American and lower socioeconomic (SES) groups. Unlike many other health risk behaviors, tobacco-related health disparities are increasing despite a large treatment network of free telephone and in-person counseling services, perhaps due to significant disparities in treatment outcomes. The goal of this project is to revise the standard treatment for tobacco dependence to address key factors associated with treatment outcome disparities and more fully meet the needs of lower SES and African American smokers thereby reducing socioeconomic disparities in tobacco dependence treatment outcomes, halting the alarming increase in tobacco-related health disparities, and reducing a leading cause of racial and socioeconomic health disparities in the US.

DETAILED DESCRIPTION:
This study will be conducted in five phases. Each phase utilizes the results from the previous phase. Each phase is also associated with at least one specific aim.

Phase One (Aim One): Complete a revised version of a standard, widely utilized, multi-component, cognitive-behavior treatment manual for tobacco dependence to include commonly utilized, cognitive-behavioral interventions that specifically address the key factors associated with treatment outcome disparities.

Phase Two (Aim Two): Using the PEN-3 Model,1-3 target and tailor RITCh_1 to address the needs of smokers who are of lower SES as well as smokers who are minority, particularly African American. In this preparatory activity, the research team will tailor and target RITCh_1 using this well-accepted theoretical model and produce the second draft of the revised treatment, called RITCh_2. Human subjects are not involved with this phase of the research. No data will be collected.

Phase Three (Aim Three): Pilot test RITCh_2 with three treatment groups (5-10 participants per group) to assess understandability and acceptability and to ensure that it can be delivered in the same 60-minute per session time frame as the standard treatment. This is a qualitative study in which the investigators will pilot test RITCh_2 with 21 participants who will be consented as pilot study participants. See Pilot Study Informed Consent Form. Contact and demographic information will be collected from participants, but not baseline and outcome assessments. Participant feedback will be provided in a group format and will not be linked to identifying information. The research team will incorporate participant feedback into a third draft of the revised treatment, RITCh_3.

Phase Four (Aim Four): Compare the effects of SES on treatment outcomes in a socioeconomically and racially diverse group of participants treated with RITCh_3 and the standard treatment. The investigators will conduct a randomized controlled trial (n=253) comparing the efficacy of RITCh_3 to the standard treatment. Investigators will use a randomized treatment design and two methods for assessing abstinence (latency to relapse and six-month point prevalence abstinence rates) to compare the effects of SES and treatment condition on treatment outcomes. Investigators expect RITCh_3 to demonstrate fewer treatment outcome disparities than standard treatment.

Phase Five (Aim Five): Compare the effects of RITCH_3 and standard treatment on each of the key factors associated with treatment outcome disparities (see Aim One and Table 1). Using analysis of covariance and logistic regression as appropriate, investigators will analyze the effects of treatment condition on each of the key factors (see Table 1). The investigators expect participants treated with RITCh_3 to demonstrate more improvement on each of the key factors than participants treated with standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* smoking cigarettes daily
* expressing a desire to quit smoking in the next 30 days
* no regular use of other tobacco products
* age 18 years or older
* no plans to move from the area in the next six months
* willing to comply with treatment
* able to engage in treatment

Exclusion Criteria:

* any contra-indication for use of the nicotine patch (i.e., uncontrolled high blood pressure, allergic reaction to patch adhesive, pregnancy, etc.),
* currently using mediations for smoking cessation (bupropion, varenicline, or any form of NRT)
* drinking more than 20 alcoholic drinks per week
* positive test on a urine screen for drugs of abuse at baseline (amphetamine, methamphetamine, cannabis, cocaine, opioids, methadone, etc.)
* current diagnosis that would prohibit engagement in brief CBT (active psychotic disorder, acute major depressive episode, significantly cognitively impaired)
* current regular use of other forms of tobacco other than smoking cigarettes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Latency to Relapse | 6 months following scheduled week 3 quit date
  Abstinence will be assessed with latency to relapse (days from Quit Date to relapse or 7 consecutive days of smoking after a 24 hour quit attempt)

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Sheffer, PhD, Principal Investigator — CCNY
Locations (1):
- The City College of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lunden SE, Pittman JC, Prashad N, Malhotra R, Sheffer CE. Cognitive, Behavioral, and Situational Influences on Relapse to Smoking After Group Treatment for Tobacco Dependence. Front Psychol. 2019 Jan 30;9:2756. doi: 10.3389/fpsyg.2018.02756. eCollection 2018. PMID 30761059